CLINICAL TRIAL: NCT06116929
Title: Functional and Cognitive Assessment of Patients With Hodgkin's Disease Undergoing Chemotherapy Before 40 Years
Brief Title: Hodgkin's Disease and Chemotherapy Before 40 Years
Acronym: FunC-AHOD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC-P00118
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hodgkin Disease
Keywords: Hodgkin Disease; Chemotherapy; Functional and Cognitive Assessment
MeSH Terms: conditions — Hodgkin Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Hodgkin's disease (Other)
  Interventions: Other: Morphological and functional magnetic resonance imaging (MRI); Other: Neuropsychological assessment
- Controls without Hodgkin's disease (Other)
  Interventions: Other: Morphological and functional magnetic resonance imaging (MRI); Other: Neuropsychological assessment

INTERVENTIONS:
Other: Morphological and functional magnetic resonance imaging (MRI) — Patients will undergo 3 morphological and functional MRI scans (during rest and activity) on the 3T MRI scanner at St Philibert Hospital (Lille, France) at 0 (M0), 6 (M6) and 12 (M12) months.
  The controls will perform a single functional MRI on the 3T MRI.
Other: Neuropsychological assessment — 3 neuropsychological assessments will be carried out at M0, M6 and M12, by the same neuropsychologist for all patients included.
  Controls will undergo the same neuropsychological assessments, but only once.

SUMMARY:
A few studies have focused on other solid cancers (colorectal, prostate). On the other hand, the study of cognitive impairment in Hodgkin's disease remains less developed, and structural and functional post-therapy MRI studies have never been carried out. The impact of cognitive impairment on Hodgkin's disease is rarely, if ever, assessed in routine clinical practice, despite the fact that it is truly disabling in 16 to 30% of patients. Cognitive impairment can persist long after diagnosis and treatment. A recent study examining cognitive functioning in patients an average of 13 years after treatment found that disorders persisted in 52% of cases, with attentional, working memory and dysexecutive (planning) difficulties. These disorders have a significant impact on the daily and professional lives of these young, often working patients. Their rapid development and persistence after treatment can therefore represent a real limiting factor, impacting both professional integration and quality of life. Finally, the current state of knowledge does not allow us to dissociate cognitive disorders from emotional disorders and fatigue, which represent a major patient complaint. A better definition of the nature, pathophysiology and specificity of these disorders would therefore enable us to take better account of their repercussions (social, professional and on quality of life) and provide better care (in terms of cognitive remediation or psychological support).

A prospective, longitudinal, multicenter, case-control interventional study in which cases are patients with Hodgkin's disease (HD) treated with CT +/- radiotherapy and controls are healthy participants will be conducted. The aim is to study the prevalence and nature of treatment-induced cognitive impairment and its correlation with emotional comorbidities, as well as structural and functional brain disorders on MRI. The patient will thus be his or her own witness, the reference state being that at the time of diagnosis, before any treatment. The fact that this state has not already been altered by the disease itself, will be verify thanks to comparison with controls.

DETAILED DESCRIPTION:
Hodgkin's disease is a neoplasia of lymphoid tissue characterized by the characteristic presence of Reed Sternberg cells. This disease is preferentially affecting young patients under the age of 40. It is the leading cause of solid cancer in adolescents and young adults. At the time of diagnosis, positron emission tomography (PET scan) is used to determine the stage of the disease. The Ann Arbor classification differentiates between localized (I-II) and disseminated (III-IV) stages. At St Vincent de Paul Hospital (Lille, France), 60-70% of diagnoses are performed at a localized stage, versus 30-40% at a disseminated stage.

Treatment is based on chemotherapy alone (disseminated forms) or a combination of chemotherapy and radiotherapy (localized forms). The average duration of treatment is around 5 months for localized forms, and between 6 and 7 months for disseminated forms. The prognosis is favorable, with a sustained complete remission rate of up to 85% in patients of all stages. The aim of treatment for these patients is therefore to achieve complete remission while reducing medium- and long-term side-effects, which could improve their quality of life.

Recently, treatment strategies have evolved, with de-escalation of chemotherapy intensity, and strategies guided by early response to Positron emission tomography (PET) scan have become the norm, in order to significantly reduce the risk of long-term side effects.

The onset of cognitive and mood disorders in patients undergoing neoplastic treatment, particularly after chemotherapy, is a frequent and disabling complication. Numerous studies have identified the occurrence of subjective and objective attentional, memory and executive disorders. However, these studies are often limited by their small size, the variability of populations, their heterogeneous design, and the variability of neuropsychological measures and criteria for defining a cognitive deficit. Furthermore, the majority of studies have focused on patients treated with chemotherapy (CT) for breast neoplasia, through neuropsychological assessment and exploration by structural and functional medical imaging. Thus, the onset of cognitive disorders (more of a dysexecutive nature) in these patients has been clearly identified, both early at the end of treatment and over the long term.

Moreover, the social, occupational and quality-of-life repercussions of these disorders have only recently been explored. However, initial results point to a positive correlation between subjective perception of cognitive functioning and quality of life. Nevertheless, the probably multifactorial etiology of these disorders remains unclear. A recent review of the literature clarifies the factors predisposing to the development of these cognitive disorders. Factors such as age and genetic polymorphisms in apolipoprotein E, catechol-O-methyltransferase and Brain-derived neurotrophic factor (BDNF) may predispose individuals to a higher risk of cognitive disorders. In addition, changes in brain morphology (reduced grey matter volume) and changes in brain connectivity could be at the root of these disorders.

In these studies, magnetic resonance imaging (MRI) identified the presence of frontal and posterior parietal gray matter volume loss in these patients. MRI also provides information on the structural and functional functioning of brain networks. For example, changes in the integrity of substance bundles have been identified using the diffusion tensor technique. In functional MRI (fMRI (BOLD signal)), numerous disturbances have been identified: hypoactivation of the prefrontal cortex and parietal lobes during activation of the executive control network, hypoactivation of the prefrontal cortex and hippocampi during tasks involving working memory, alteration of the dorsal attentional network and the default mode network.

In addition, one study suggests the presence of pre-treatment network alterations in patients with breast neoplasia. At pathophysiological level, animal models suggest the involvement of alterations in neurogenesis, mitochondrial dysfunction or cerebral cytokine response.

ELIGIBILITY:
Inclusion criteria - case :

* Patient with newly diagnosed Hodgkin's disease
* With intention to treat with chemotherapy +/- radiotherapy
* Aged between 18 and 40 years
* Fluency in French
* Able to undergo neuropsychological evaluation (absence of major sensory disorders)
* Agreeing to take part in the study and having signed the informed consent form
* Affiliated with a social security scheme

Inclusion criteria - controls:

* Individual without Hodgkin's disease
* Aged between 18 and 40
* Proficient in French
* Agreeing to participate in the study and having signed the informed consent form
* Affiliated with a social security scheme

Cases and controls will be matched on age (± 5 years difference), and number of years of education (difference ≤ 2 years).

Non-inclusion criteria - cases + controls :

* Claustrophobia preventing MRI from being performed
* Contraindication to MRI
* Previous chemotherapy
* History of neurological or psychiatric illness, including severe depression, or cognitive impairment
* Use of medications that may cause neurological or psychiatric signs
* Alcohol or drug abuse
* Pregnant women
* Persons under guardianship or trusteeship

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Computerized Speed Cognitive Test (CSCT) | 12 months
  The CSCT will be used to evaluate the impact of Chemotherapy +/- radiotherapy treatment on the attentional abilities of HD cases, immediately after the end of treatment, and at a distance from this treatment.
  The CSCT score is calculated as follows:
  The patient has 90 seconds to orally state the correspondence of numbers (from 1 to 9) to 9 different symbols (matched according to a correspondence standard). The number of correct answers is measured (maximum score of 120).

SECONDARY OUTCOMES:
Brief Visual-spatial Memory Test-Revised | 12 months
  Recall performance is recorded for each of the immediate recall trials (Trial 1, Trail 2, and Trial 3) and for the delayed recall trial (Delayed Recall).
  The recall scores are combined to form three additional summary measures of learning and memory.
  Recognition Hits and False Alarms are recorded during the delayed recognition task. Recognition Hits are calculated as the number of correct "YES" responses to target items, and Recognition False Alarms are calculated as the number of incorrect "yes" responses to nontarget items.
D2-R | 12 months
  The d2-R tests the candidate's ability to discriminate details in a short space of time, while maintaining concentration. Candidates must locate and cross out target characters (d with 2 lines) from a large number of distractors in less than 20 seconds for each series.the candidate's index reflects his or her performance compared to people in his or her age group. A European sample of over 2,100 subjects aged between 18 and 55, representative of the population, is used as a reference.
Trail Making test | 12 months
  The Trail Making Test (TMT) is a freely available, timed, neuropsychological test that involves visual scanning and working memory. The TMT has two parts; the TMT-A (rote memory) and TMT-B (executive functioning).85 In each test the participant is asked to draw a line between 24 consecutive circles that are randomly arranged on a page. The TMT-A uses all numbers, whereas the TMT-B alternates numbers and letters, requiring the patient to switch between numbers and letters in consecutive order. The TMT is scored by how long it takes to complete the test. The time includes correction of errors prompted by the examiner. If the person cannot complete the test in 5 minutes, the test is discontinued. An average score for TMT-A is 29 seconds and a deficient score is greater than 78 seconds. For TMT-B, an average score is 75 seconds and a deficient score is greater than 273 seconds.
Functional Assessment of Cancer Therapy- Cognitive Function (FACT-Cog) | 12 months
  The FACT-Cog is a 37-item self-response measure to assess cognitive concerns of cancer patients, consisting of four subscales. The patient indicates how often the situation occurred during the last 7 days, on a 5-point Likert scale ("0 = Never" to "4 = Several times a day").
Hospital Anxiety and Depression scale (HAD) | 12 months
  The HAD scale i comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven to depression (total D), giving two scores (maximum score for each = 21).To screen for anxiety and depressive symptoms, the following interpretation:
  To screen for anxiety and depressive symptoms, the following :
  * 7 or less: no symptoms
  * 8 to 10: doubtful symptomatology - 11 or more: symptomatology.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | 12 months
  The Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) is a 13-item measure that assesses self-reported fatigue and its impact upon daily activities and function. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued)
Impact on Participation and Autonomy (IPA) scale | 12 months
  The IPA quantifies limitations in participation and autonomy. To this extent it contains 32 items. Each of these 32 items has identical response options, ranging from zero to four with higher scores representing poorer participation and autonomy:
  Response options (scoring):
  0 Very good
  1. Good
  2. Fair
  3. Poor
  4. Very poor
Marshall test | 12 months
  This test is based on two questions:
  (A) How many times a week, do you usually do 20 minutes of vigorous physical activity that makes you sweat or puff and pant? (for example, jogging, heavy lifting, digging, aerobics, or fast bicycling) N .3 times/week N 1-2 times/week N none
  Score:
  N 4 N 2 N 0 (B) How many times a week, do you usually do 30 minutes of moderate physical activity or walking that increases your heart rate or makes you breath harder than normal? (for example, mowing the lawn, carrying light loads, bicycling at a regular pace, or playing doubles tennis) N . 5 times/week N 3-4 times/week N 1-2 times/week N none
  Score:
  N 4 N 2 N 1 N 0 Total: score A + score B Score >4 = ''Sufficiently'' active Score 0-3 = ''Insufficiently'' active

CONTACTS AND LOCATIONS:
Overall Officials: Sandy AMORIM, Principal Investigator — Onco-Hematology Department-Hôpital Saint Vincent de Paul-GHICL
Locations (4):
- France (4):
  - Centre Hospitalier Artois Ternois, Arras
  - Hôpital Claude Huriez, Lille
  - Hôpital Saint-Philibert, Lomme
  - Hôpital Victor Provo, Roubaix

IPD SHARING:
Plan to Share IPD: No